CLINICAL TRIAL: NCT04872270
Title: Multimodal Postoperative Pain Management Following Shoulder Arthroplasty
Brief Title: Pain Management After Shoulder Arthroplasty
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FTJO21D.060
Record Dates: First submitted 2021-05-03; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Caffeine; Pain, Joint
MeSH Terms: conditions — Arthralgia | interventions — Arthroplasty, Replacement, Shoulder; Caffeine; oxycodone-acetaminophen; Ondansetron; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Caffeine Group (Active Comparator): 2 week supply of 100mg caffeine + aspirin 325mg + standard pain regimen (experimental)
  Interventions: Procedure: Total Shoulder Arthroplasty; Drug: Caffeine Pill; Drug: Percocet 10Mg-325Mg Tablet; Drug: Zofran 4Mg Tablet
- No Caffeine Group (Active Comparator): aspirin 325mg + standard pain (control)
  Interventions: Procedure: Total Shoulder Arthroplasty; Drug: Percocet 10Mg-325Mg Tablet; Drug: Zofran 4Mg Tablet

INTERVENTIONS:
Procedure: Total Shoulder Arthroplasty — Participant will have total shoulder replacement
Drug: Caffeine Pill — 2 week supply of 1000 mg caffeine given postoperatively as part of the pain regimen
  Arms: Caffeine Group
Drug: Percocet 10Mg-325Mg Tablet — given postoperatively as standard post-op pain management
Drug: Zofran 4Mg Tablet — given postoperatively as standard post-op management

SUMMARY:
Pain control is a critical after many surgical procedures. It is well known that orthopaedic surgeries are among the most painful procedures, with total joint arthroplasty being a clear example of this situation. Current trends in pain management are morphing and multimodal opioid sparing protocols are now being evaluated and implemented, with results showing a decrease in the amount of opioids being prescribed. Despite all efforts, most patients experience pain and, in order to control it, multiple medications have been tried with variable results. The most commonly prescribed medications are opioids, but side effects associated with their use as well as their addictive potential are making them a less desirable option for patients. Currently there is a trend towards diminishing opioids consumption and prescribing alternative pain control regimens.Caffeine is a well known molecule that when associated with non-steroidal anti-inflammatory drugs (NSAIDS) potentiates their analgesic effect and decreases the amount of doses required to control pain. Little is known about the effect of caffeine over pain relief in patients undergoing total joint arthroplasty, but preliminary results in other fields make us believe it could have a potential benefit for patients undergoing total joint arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who undergo primary Total Shoulder Arthroplasty or Reverse Total Shoulder Arthroplasty
* Patient willing and able to complete postoperative surveys
* Post-Menopausal Women and Men over the age of 55

Exclusion Criteria:

* Patients reporting caffeine consumption in excess of 300mg daily
* Patient has known history of opioid addiction, has taken opioids preoperatively, or other forms of substance abuse.
* Patient has history of cardiac diseases that might be aggravated by the use of caffeine, as diagnosed by a cardiologist or demonstrated by an abnormal EKG.
* Patient has a known allergy to aspirin or caffeine.
* Patient has history of cancer, neuropathic pain, or nerve degenerative disease that would affect patient reported outcomes including pain.
* Patient has history of anxiety disorder
* Patients with known sleep disturbances that would otherwise be affected by caffeine
* Patients undergoing revision surgery
* Patients who require alternate DVT prophylaxis other than ASA.
* Patients undergoing inpatient arthroplasty
* Workman's comp patient or patient has current litigation pending

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
postoperative shoulder function | 24 weeks
  This will be measured using the Simple Shoulder Test (SST) which consist of 12 questions
Postoperative shoulder function | 24 weeks
  This will be measured using the American Shoulder and Elbow Surgeon Survey (ASES)
Postoperative Pain | 15 days
  This will be measured using the Visual Analog Scale for Pain (VAS) survey

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States